CLINICAL TRIAL: NCT02273284
Title: Pain Perception of Children and Youth Receiving Non-sedated Botulinum Toxin-A Injections Using the Buzzy®
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: we identified that the device tested in this study was not approved by Health canada
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Ronit Mesterman, Pediatric Neurologist, Associate professor of Pediatrics, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no number yet
Record Dates: First submitted 2014-10-19; First posted 2014-10-23 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: Pain, Pediatrics, Botulinum Toxin injections, Buzzy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buzzy (Experimental): Participants will use the Buzzy, a small vibration device during their Botulinum toxin treatments. The Buzzy will be held over the injection site for 30 sec prior to the injection, then will be moved more rostral during the actual injection. The Buzzy will be applied in the same fashion to each targeted muscle.
  Interventions: Device: Buzzy
- control - no Buzzy (No Intervention): Participants in the control group will receive their regular Botulinum toxin treatment without the use of the Buzzy

INTERVENTIONS:
Device: Buzzy — The Buzzy will be applied for 30 seconds over the area that is going to be injected, then during the actual injection the Buzzy will be moved rostrally and continuously used during the injection. When the injection is completed the Buzzy is positioned in the same way over the next injection site.
  Other Names: vibration therapy
  Arms: Buzzy

SUMMARY:
The use of Botulinum toxin injections (BoNT-A) has become a standard therapy for children and youth who suffer from stiffness of their muscles due to a neurological problem. These injections are given into each muscles which require treatment, which often means receiving multiple injections in one session. Intramuscular injections are typically painful. Treatment can be provided unsedated and then should incorporate distraction and relaxation techniques, or can be alternatively be provided with the use of sedation.

To improve the pain experience the investigators want to assess the feasibility and impact on the pain perception when using a vibration device called the Buzzy during BoNT-A injections. The Buzzy creates a vibration that is applied over the injection site for 30 seconds before the injection and will be continued just above the injection site during the injection. The Buzzy has been shown to help reduce pain in procedures such as i.v. insertions and immunizations, but has not been tested in children and youth receiving multiple BoNT-A injections.

DETAILED DESCRIPTION:
Children and youth who receive hypertonia treatment with non-sedated BoNT-A injection will be invited to participate in this clinical trial. The patients will be randomized to receiving the injection with the Buzzy versus the control group without the Buzzy. Both groups will still receive their typical supports that will include their choice of local anesthetic cream, relaxation and distraction techniques. Randomization will be stratified for the ability to self report.

Measures to capture the pain will include self report of pain, by using the Face Pain Scale revised (FPSr) in all participants who are able to self report. In addition all participants will be evaluated by the use of the Face, Legs, Activity, Cry and Consolability scale (FLACC scale), an observational tool validated to capture pain responses. The investigators will also include measurement of heart rate at rest, during and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any child and youth who receives non-sedated Botulinum toxin-A injections and is interested and consenting to using the Buzzy

Exclusion Criteria:

* Patients receiving Botulinum Toxin-A injections under sedation
* Patients younger than 2 years or older than 18 years.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale revised | The participants will be asked to rate their pain 3 minutes after the treatment. This will take about 2-5 minutes.
  pain will be assessed by the use of the FPSr, a tool which was validated and been shown to be reliable in children and youth age 4 years and up.

SECONDARY OUTCOMES:
FLACC scale (base line) | Baseline: Participants will be observed and rated on the FLACC scale 1 minute prior to the intervention.
  The FLACC scale is a validated observational measure to rate bodily responses to pain. The scale has five items. Each item observes one area/activity and includes the following: face, legs, activity, cry and consolability. Each item can get a score of 0 (no response) to 2 (most response) so that the total FLACC score can vary from 0-10.
FLACC scale (during intervention) | Participants will be observed and rated on the FLACC scale during the intervention. Intervention time is typically 1-3 minutes.
  The FLACC scale is a validated observational measure to rate bodily responses to pain. The scale has five items. Each item observes one area/activity and includes the following: face, legs, activity, cry and consolability. Each item can get a score of 0 (no response) to 2 (most response) so that the total FLACC score can vary from 0-10.
FLACC scale (after intervention) | Participants will be observed and rated on the FLACC scale 5 minutes after the intervention.
  The FLACC scale is a validated observational measure to rate bodily responses to pain. The scale has five items. Each item observes one area/activity and includes the following: face, legs, activity, cry and consolability. Each item can get a score of 0 (no response) to 2 (most response) so that the total FLACC score can vary from 0-10.
Heart rate (baseline) | The heart rate will be captured 1 minute before the intervention
  Heart rate will be measured before, during and after the intervention. Heart rate has been shown to be a biological marker of stress and pain.
Heart rate (during intervention) | The heart rate will be captured during the intervention.
  Heart rate will be measured before, during and after the intervention. Heart rate has been shown to be a biological marker of stress and pain.
Heart rate (after intervention) | The heart rate will be captured 5 minutes after the intervention.
  Heart rate will be measured before, during and after the intervention. Heart rate has been shown to be a biological marker of stress and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Mesterman, M.D., Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Lukban MB, Rosales RL, Dressler D. Effectiveness of botulinum toxin A for upper and lower limb spasticity in children with cerebral palsy: a summary of evidence. J Neural Transm (Vienna). 2009 Mar;116(3):319-31. doi: 10.1007/s00702-008-0175-8. Epub 2009 Jan 14. PMID 19142573
- [Background] Uman LS, Chambers CT, McGrath PJ, Kisely S. A systematic review of randomized controlled trials examining psychological interventions for needle-related procedural pain and distress in children and adolescents: an abbreviated cochrane review. J Pediatr Psychol. 2008 Sep;33(8):842-54. doi: 10.1093/jpepsy/jsn031. Epub 2008 Apr 2. PMID 18387963
- [Background] Moayedi M, Davis KD. Theories of pain: from specificity to gate control. J Neurophysiol. 2013 Jan;109(1):5-12. doi: 10.1152/jn.00457.2012. Epub 2012 Oct 3. PMID 23034364
- [Background] Fehlings D, Narayanan U, Andersen J, Beauchamp R, Gorter JW, Kawamura A, Kiefer G, Mason M, McCormick A, Mesterman R, Switzer L, Watt J. Botulinum toxin-A use in paediatric hypertonia: Canadian practice patterns. Can J Neurol Sci. 2012 Jul;39(4):508-15. doi: 10.1017/s0317167100014049. PMID 22728860
- [Background] Whelan HM, Kunselman AR, Thomas NJ, Moore J, Tamburro RF. The impact of a locally applied vibrating device on outpatient venipuncture in children. Clin Pediatr (Phila). 2014 Oct;53(12):1189-95. doi: 10.1177/0009922814538494. Epub 2014 Jun 12. PMID 24924565
- [Background] Canbulat N, Ayhan F, Inal S. Effectiveness of external cold and vibration for procedural pain relief during peripheral intravenous cannulation in pediatric patients. Pain Manag Nurs. 2015 Feb;16(1):33-9. doi: 10.1016/j.pmn.2014.03.003. Epub 2014 Jun 7. PMID 24912740
- [Background] Sharma P, Czyz CN, Wulc AE. Investigating the efficacy of vibration anesthesia to reduce pain from cosmetic botulinum toxin injections. Aesthet Surg J. 2011 Nov;31(8):966-71. doi: 10.1177/1090820X11422809. Epub 2011 Oct 14. PMID 22001341
- [Background] Russell K, Nicholson R, Naidu R. Reducing the pain of intramuscular benzathine penicillin injections in the rheumatic fever population of Counties Manukau District Health Board. J Paediatr Child Health. 2014 Feb;50(2):112-7. doi: 10.1111/jpc.12400. Epub 2013 Oct 18. PMID 24134180
- [Background] Roy EA, Hollins M, Maixner W. Reduction of TMD pain by high-frequency vibration: a spatial and temporal analysis. Pain. 2003 Feb;101(3):267-274. doi: 10.1016/S0304-3959(02)00332-9. PMID 12583869
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Koenig J, Jarczok MN, Ellis RJ, Hillecke TK, Thayer JF. Heart rate variability and experimentally induced pain in healthy adults: a systematic review. Eur J Pain. 2014 Mar;18(3):301-14. doi: 10.1002/j.1532-2149.2013.00379.x. Epub 2013 Aug 6. PMID 23922336